CLINICAL TRIAL: NCT05638191
Title: Nerve Transfer Surgery to Restore Upper-limb Function After Ceervical Spinal Cord Injury
Brief Title: Nerve Transfer Surgery to Restore Upper-limb Function After Cervical Spinal Cord Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Queen's University (Other); Dalhousie University (Other); University of Toronto (Other); Wings for Life (Other)
Responsible Party: Principal Investigator, Michael Berger, Clinical Assistant Professor, University of British Columbia
Other Study IDs: H20-03350
Record Dates: First submitted 2022-11-01; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Spinal Cord Injury; Spinal Cord Injury at C5-C7 Level; SCI - Spinal Cord Injury; Upper Extremity Paralysis; Upper Extremity Dysfunction; Tetraplegia; Upper Extremity Paresis; Cervical Spinal Cord Injury
Keywords: spinal cord injury; upper extremity nerve transfer; nerve transfer; SCI; nerve reconstruction; quadriplegia; paresis
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia; Paresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experiemental: Surgical Arm: Individuals in this group will receive nerve transfer surgery 6 - 9 months post cervical spine injury and be observed for two years post-operatively.
- Control: Non-surgical: Individuals in this group will not have undergone nerve transfer surgery. They will be observed for two years post injury while receiving standard of care including medical and rehabilitation. We want to reinforce that individuals are not being randomized to surgery versus non-surgery. Rather individuals this group will either have made the decision not to undergo surgery, independent their participation in this study.

SUMMARY:
The goal of this prospective, open label cohort study is to assess functional and motor outcomes in individuals with cervical spinal cord injury who have undergone nerve transfer surgery, with the goal of increasing upper limb function. We will also compare these outcomes to a cohort of similarly matched individuals who have not undergone nerve transfer surgery, using robust outcome measures, rigorous pre-operative clinical and neurophysiological assessments, and standardized rehabilitation. At the end of this project we aim to develop a model for predicting nerve transfer outcomes using pre-operative clinical and neurophysiological characteristics.

DETAILED DESCRIPTION:
The purposes of this study are:

1. To quantify functional and motor outcomes of NT in patients with SCI, using robust outcome measures, rigorous pre-operative clinical and neurophysiological assessments, and standardized rehabilitation, and to compare these outcomes against individuals who did not undergo nerve transfer surgery.
2. To develop a model for predicting NT outcomes using pre-operative clinical and neurophysiological characteristics.

Outcome measures:

Purpose 1: The primary study outcome is the Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP Ver. 1). Secondary outcomes are the Spinal Cord Independence Measure (SCIM) and motor outcomes in recipient muscles following NT, including muscle strength and neurophysiological assessments at 3 months intervals post-operatively, to final outcome measurement at 24 months.

Purpose 2: Relevant demographic, clinical variables and neurophysiological variables (including joint range of motion, muscle spasticity, pain, depression motor unit number estimation in recipient muscles and ultrasound evaluation of recipient muscle quality), are a priori variables that will be collected at baseline, in order to develop a clinical prediction tool to inform prognosis.

Research Design:

All SCI individuals referred to an interdisciplinary clinic for potential nerve transfer will undergo a standardized clinical examination, according to the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI), to classify neurological level of injury. As well, electrodiagnostic test which will be performed by one of our highly qualified physicians. Individuals who are deemed candidates for nerve transfer surgery will be screened and invited to participate in the study. Participation in the study will not, in any way, influence clinical care.

After receiving written consent, outcome measurement will take place pre-operatively, then at 3-month intervals post operatively; final analysis will occur at 24 months after surgery. As well, a control group consisting of those SCI individuals who chose to not undergo or are not candidates for surgery will be recruited. This "control group" will undergo assessments at 24 months following their injuries, in line with the anticipated functional plateau in spontaneous recovery expected . Outcome measurement will be performed at GF Strong Rehabilitation Hospital (Primary site), the International Collaboration on Repair Discoveries (ICORD), Sunnybrook Hospital in Toronto, and Kingston Health Science Centre. Rehabilitation will be administered by highly qualified hand therapists with standardized frequency, and duration for all individuals. All study data will be stored in a REDCap database which will be shared between all participating institutions.

Outcome measurement & information collected include:

Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP), which is a validated upper limb functional measure, specifically designed for use in SCI (Kalsi-Ryan et al. 2012). It incorporates three domains vital to upper limb function: sensation, strength, and prehension. It is a multimodal test comprising 5 subtests for each upper limb: dorsal sensation, palmar sensation, strength, prehension ability and prehension performance. The GRASSP results in 5 numerical scores that provide a comprehensive profile of upper-limb function and will be administered by GRASSP certified research personnel. As well, individuals will be asked to complete the Spinal Cord Independence Measure (SCIM) questionnaire (Catz A, et al. 1997) on the same day of their visit.

At Baseline, a validated technique called motor unit number estimation (MUNE) counts the number of MN's and can be essential in evaluating MN health. We aim to carry out this technique towards measuring the health of MN's in functionally relevant muscles in patients with SCI and comparing this with healthy controls. The purpose of this study is to provide a quantitative measure of the size of MN pool in clinically relevant muscles below the level of SCI using MPS and MScan MUNE. We will also supplement information about MNs with ultrasound-derived measures of muscle quality.

Ultrasound sonography recording will be taken to analyze the structural health of recipient muscles and to quantify muscle fibrosis and atrophy. The muscles of interest will be anatomically identified and marked, and ultrasound gel will be applied to skin surface of the upper limb prior to placing the ultrasound probe. Individuals will be asked to lie in a dimly lit room for this portion of the study.

Demographic information will be collected for each participant, including

* age;
* sex;
* medical comorbidities; and
* medications

Clinical factors influencing functional and motor recovery in SCI will be measured:

* spasticity with modified Ashworth scores;
* depression with Beck's depression inventory (Beck, A. T., et al. 1996);
* passive ranges of motion in joints targeted by NT; and
* brief pain inventory (Ullrich PM, et al. 2008).

ELIGIBILITY:
Inclusion Criteria:

* Motor complete (AIS A or B) between neurological level of injury C5 and C8
* Able to provide informed written consent
* Able to attend and comply with the testing protocols
* Able to understand and speak English or have access to an appropriate interpreter as judged by the investigator.

Exclusion Criteria:

* An uncontrolled medical condition (e.g. uncontrolled cardiovascular disease, diabetes, kidney or liver disease)
* Have ever received botulinum toxin injections (Botox) for tone management in the upper limb
* An unmanaged secondary complication of SCI including but not limited to uncontrolled neuropathic pain or spasticity, syringomyelia, fracture, urinary tract infection or significant pressure ulcer, preventing participation in testing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient referrals are ensured through established care pathways for upper-limb rehabilitation in SCI, including nerve transfer. Research objectives will be facilitated through already available institutional clinical and rehabilitation resources at each study site. Potential participants will be informed of the study directly by their treating physicians. The research study will be introduced by the PI or one of the co-Is of the study, who are also responsible for clinical care of all prospective participants.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-06-03 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) | Baseline then every 3 months for 2 years
  A validated upper limb functional measures and previously is used in SCI (Kalsi-Ryan et al. 2012) incorporates three domains vital to upper limb function: sensation, strength, and prehension.

SECONDARY OUTCOMES:
Modified Ashworth scores (MAS) | Baseline then every 3 months for 2 years
  Modified Ashworth Scale (MAS) have been utilized in spinal cord injury patient population to assess spasticity by examining muscle tones.
Range of Motion | Baseline then every 3 months for 2 years
  A Goniometer is used to measure range of motion of the joint angles (degrees) from the axis of the joint. The measurement of joint movements is compared to its full potential.
Ultrasound | Baseline then every 3 months for 2 years
  Ultrasound imaging to assess the structural health of recipient muscles and to quantify muscle fibrosis and atrophy.
Spinal Cord Independence Measure (SCIM) | Baseline then every 3 months for 2 years
  The SCIM has been developed to address three specific areas of function in patients with spinal cord injuries such as activities of daily living, respiration and sphincter management, and a patient's mobility abilities.
Douleur Neuropathique 4 (DN-4) | Baseline then every 3 months for 2 years
  A questionnaire consisting of 10 items and can be useful in assessment of neuropathic pain. The items related to pain quality are based on an interview and examination of the patient.
Beck's Depression Inventory (BDI) | Baseline then every 3 months for 2 years
  The questionnaire is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Berger, MD, PHD, Principal Investigator — University of British Columbia
Locations (4):
- Canada (4):
  - GF Strong Rehabilitation Hospital, Vancouver, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided
The IPD sharing plan is under discussion.